CLINICAL TRIAL: NCT05896579
Title: Identifying Patterns of Resting and Exertional Right Ventricular Dysfunction Among Patients With Chronic Obstructive Pulmonary Disease and Pulmonary Artery Enlargement
Brief Title: Identifying Right Ventricular Dysfunction in COPD Through Right Heart Catheterization, Imaging and Exercise
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 23-0516
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2024-08-09 (Actual); Status verified 2024-08

CONDITIONS: COPD; Pulmonary Hypertension; Right Ventricular Dysfunction
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Hypertension, Pulmonary; Ventricular Dysfunction, Right | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Study participants will undergo testing to identify patterns of right ventricular dysfunction. If a study participant decides to participate in exercise training, the participant will complete an exercise training intervention followed by repeat testing to determine impact of exercise training on right ventricular dysfunction.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- COPD with pulmonary artery enlargement (Experimental): Participants will complete testing at rest and during exercise to identify patterns of right ventricular dysfunction. If a participant decides to participate in the optional exercise training program, the participant will complete exercise training followed by repeat testing to determine the impact of exercise training on right ventricular dysfunction.
  Interventions: Behavioral: Exercise training

INTERVENTIONS:
Behavioral: Exercise training — Exercise training will include supervised high-intensity interval training for ~35 minutes 3x/week on an upright stationary bicycle and unsupervised continuous aerobic exercise for ~30 minutes 2x/week.

SUMMARY:
This study plans to learn more about heart function among individuals with chronic obstructive pulmonary disease (COPD). In particular, the investigators want to understand the different patterns of right ventricular response to pulmonary hypertension (high pressure in the lungs) during rest and exercise. By identifying patterns of right ventricular dysfunction, this study will help identify better treatments for patients with COPD in the future.

ELIGIBILITY:
Inclusion Criteria:

* COPD (determined by ratio of forced expiratory volume in 1 second to forced vital capacity [FEV1/FVC] <0.7) • Pulmonary artery enlargement determined by pulmonary artery-to-aorta ratio >1 or >30 mm on most recent CT

Exclusion Criteria:

* Exacerbation of COPD or use of systemic corticosteroids in the 3 months prior to enrollment
* Change in COPD therapy in the 3 weeks prior to enrollment
* Requirement of >6 LPM supplemental oxygen at rest
* Requirement of >10 LPM with exertion
* Active/uncontrolled cardiovascular disease (e.g. hypertension with blood pressure >150/100 despite antihypertensives; coronary artery disease with angina; left ventricular ejection fraction ≤40%; arrhythmia; pulmonic, mitral or aortic valvular abnormality greater than mildin severity; tricuspid regurgitation greater than moderate in severity; diabetes with HbA1c >8.5%)
* Volume overload (jugular vascular distension or greater than trace peripheral edema)
* Interstitial lung disease
* Untreated severe obstructive sleep apnea
* Active malignancy
* Medical conditions that limit exercise on an upright stationary bicycle (e.g. osteoarthritis, etc.)
* Pregnancy
* Body mass index <18 or >35
* Hematocrit <25% or >55%
* For optional Part 2 i.e. exercise training and Visit 2, residence >90 miles from University of Colorado Anschutz Medical Campus or unwillingness/inability to attend exercise training sessions for approximately 35 minutes 3x/week for 12 weeks
* For optional Part 2 i.e. exercise training and Visit 2, already engaged in routine exercise training (>30 minutes at >3 METs 3 times/week or more)

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2023-08-22 (Actual); Primary Completion 2030-07 (Estimated); Study Completion 2030-07 (Estimated)

PRIMARY OUTCOMES:
Right ventricular-arterial coupling measured by conductance catheter | Up to 1 hour
  Ratio of end-systolic elastance to effective arterial elastance (Ees/EA)

SECONDARY OUTCOMES:
Mean pulmonary artery pressure measured by pulmonary artery catheter | Up to 1 hour
  In mmHg
Cardiac output measured by pulmonary artery catheter | Up to 1 hour
  In L/min, calculated by Fick equation
Right ventricular contractility measured by conductance catheter | Up to 1 hour
  Maximum rate of pressure change, dP/dtmax in mmHg/sec
Right ventricular lusitropy measured by conductance catheter | Up to 1 hour
  Minimum rate of pressure change, dP/dtmin in mmHg/sec
Right ventricular energetics, measured by conductance catheter | Up to 1 hour
  Stroke work in mmHg*mL
Maximum oxygen consumption (VO2max) | Up to 1 hour
  In L/min
Red blood cell acylcarnitine 10:0 measured by peripheral venous metabolomics(ultra-high performance liquid chromatography coupled to mass spectrometry) | Up to 1 hour
  Relative ion count
Plasma acylcarnitine 10:0 measured by peripheral venous metabolomics (ultra-high performance liquid chromatography coupled to mass spectrometry) | Up to 1 hour
  Relative ion count
Health-related quality of life by Short Form 36 (SF-36) questionnaire | Up to 1 hour
  Units, range 0-100 with greater scores indicating a more favorable health state
Right to left ventricle diameter ratio measured by computed tomography | Up to 1 hour
  Ratio of right ventricle diameter to left ventricle diameter
Distal pulmonary vascular pruning measured by computed tomography | Up to 1 hour
  Ratio of total volume of small pulmonary blood vessels defined by cross-sectional area <5 mm2 to total volume of all pulmonary blood vessels
Right ventricular contractility measured by transthoracic echocardiography | Up to 1 hour
  Rate of pressure change, tricuspid dP/dt in mmHg/sec
Exercise training feasibility | 4 months
  Proportion of exercise training sessions completed
Exercise training safety | 4 months
  Adverse events, reported or observed

CONTACTS AND LOCATIONS:
Overall Officials: Lindsay Forbes, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Anschutz Medical Campus, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No